CLINICAL TRIAL: NCT02230527
Title: Establishing the Microcirculatory Effects of Ticagrelor on Tissue Perfusion in Critical Limb Ischemia
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Joseph Campbell, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-799
Record Dates: First submitted 2014-08-26; First posted 2014-09-03 (Estimated); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Clopidogrel (Active Comparator): Clopidogrel 75mg by mouth daily
  Interventions: Drug: Clopidogrel
- Ticagrelor (Experimental): Ticagrelor 90mg by mouth twice daily
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — 90mg twice a day by mouth
  Other Names: Brilinta; Brilique; Possia
  Arms: Ticagrelor
Drug: Clopidogrel — 75mg once a day by mouth
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
This is a single center, prospective, randomized, unblinded, open-label, active controlled pilot study to evaluate the efficacy and safety of ticagrelor plus aspirin versus clopidogrel plus aspirin in patients with Rutherford Stage IV to VI PAD that have undergone a percutaneous transluminal angioplasty (PTA) of the lower extremities in the past 2 weeks.

DETAILED DESCRIPTION:
Enrollment into the study will require severe symptomatic CLI without wounds (Rutherford Stage IV) or CLI with concomitant vascular insufficiency wounds (Rutherford Stage V-VI PAD).

Potential participants will be identified and screened prior to discharge or at the time of the first out-patient visit (within 2 weeks after discharge) after a percutaneous lower extremity arterial angiography with arterial intervention (stent or balloon angioplasty) for the presence of lower extremity vascular insufficiency. Participants will be classified as Rutherford Class IV - VI (with or without ulcerations). A total of 60 patients will be randomized into 2 treatment groups in a 1:1 ratio (ticagrelor to clopidogrel). Patients are placed on clopidogrel after their arterial intervention per standard of care. They will remain on clopidogrel up to the time that randomization occurs. For patients that are randomized to ticagrelor, the clopidogrel will be stopped.

Patients will be randomized to either ticagrelor 90mg by mouth twice daily or clopidogrel 75mg by mouth daily.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18-100 years with Rutherford Classification Stage IV through VI PAD with a recent percutaneous lower extremity arterial angiography with arterial intervention in the past 2 weeks
2. Willingness to sign informed consent
3. Ability to return for follow up visits
4. A female patient of childbearing potential who is sexually active must agree to use adequate contraception from screening until 30 days after receiving the last dose of study drug. Women not of childbearing potential are defined as those who have surgically sterilized (hysterectomy, bilateral oophorectomy, or tubal ligation) or who are post menopausal (defined as at least 2 years since last regular menses). The female patient should not be lactating and must have a negative pregnancy test at screening.

Exclusion Criteria:

Patients will be ineligible for this study if they meet any one of the following criteria:

1. Intolerance to thienopyridines
2. Hypersensitivity to ticagrelor or any component of the product.
3. Concomitant use of oral anticoagulation with vitamin K antagonist, factor Xa inhibitor, or direct thrombin inhibitor
4. History of intracranial hemorrhage
5. History of severe hepatic impairment defined by baseline transaminase greater than or equal to 3x ULN or any elevation in bilirubin
6. Active bleeding
7. Allergy to aspirin
8. Baseline TcPO2 < 10 mmHg post angiography
9. Resting, pre- procedure heart rate <50 beats-per-minute without a permanent pacemaker and not on an atrioventricular nodal blocking agent
10. Severe COPD on home oxygen therapy -

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Campbell, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clopidogrel | Ticagrelor
Started | 23 | 23
Completed | 18 | 21
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clopidogrel | Ticagrelor | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (11.8) | 67.2 (8.9) | 66.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 13 | 18 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 11 | 15 | 26
  Asian | 1 | 0 | 1
  African American/Black | 11 | 8 | 19
Past/Current Smoker [Count of Participants; unit: Participants] | 18 | 16 | 34
History of Hypertension [Count of Participants; unit: Participants] | 20 | 20 | 40
History of Diabetes [Count of Participants; unit: Participants] | 17 | 15 | 32
History of Hyperlipidemia [Count of Participants; unit: Participants] | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in TcPO2 From Baseline to Month 6
Description: The primary endpoint is the absolute change in TcPO2 from baseline to month 6 compared between treatment groups.
Time Frame: 6 months
Population: Patients with baseline and TCPO2 data available at 6 months
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Clopidogrel | Ticagrelor
Number analyzed (Participants) | 16 | 15
mmHG | 14.9 (17.8) | 4.2 (19.9)

ADVERSE EVENTS:
Time Frame: Through 6 months
Description: Serious adverse events
Arm/Group | Clopidogrel | Ticagrelor
All-Cause Mortality (participants affected / at risk) | 1/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 5/23 | 6/23
Other Adverse Events (participants affected / at risk) | 3/23 | 9/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel (N=23) | Ticagrelor (N=23)
Worsening Limb Ischemia (Vascular disorders) | 1 (2) | 3 (3)
Limb pain/ulcer (Vascular disorders) | 2 (2) | 4 (4)
infection (Infections and infestations) | 1 (1) | 2 (2)
Organ failure (General disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Amputation (Surgical and medical procedures) | 0 (0) | 2 (2)
Stent occlusion (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel (N=23) | Ticagrelor (N=23)
UTI (Renal and urinary disorders) | 1 (1) | 0 (0)
Junctional rhythm (Cardiac disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Foot ulcer (Vascular disorders) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Excessive bruising (Vascular disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT02230527/Prot_SAP_000.pdf